CLINICAL TRIAL: NCT07218003
Title: An Open-Label, Multicenter, Phase 1/1b Study of RNDO-564 as Monotherapy and in Combination With Pembrolizumab in Adult Participants With Relapsed/Refractory Locally Advanced or Metastatic Urothelial Cancer and Other Solid Tumors Associated With Nectin-4 Expression
Brief Title: A Phase 1/1b of RNDO-564 Single Agent or in Combination With Pembrolizumab in Bladder Cancer and Other Solid Tumors Associated With Nectin-4
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rondo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RNDO-564-001
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer; Cervical Cancer; Head and Neck Squamous Cell Cancer; Triple Negative Breast Cancer (TNBC); Urothelial Carcinoma Bladder; Gastroesophageal Junction (GEJ) Adenocarcinoma; Esophageal Squamous Cell Cancer; Gastric Cancer; Cancer; Solid Tumors (Phase 1)
Keywords: RNDO-564-001; bladder cancer; bispecific antibody; solid tumors; Nectin-4; dose escalation; Phase 1/1b; CD28 x Nectin-4 bispecific; T-cell engager; CD28 costimulation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms; Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Stomach Neoplasms; Neoplasms; Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Single Agent Dose Level 1 (Experimental): Single Agent Dose Level 1
  Interventions: Drug: RNDO-564
- Single Agent Dose Level 2 (Experimental): Single Agent Dose Level 2
  Interventions: Drug: RNDO-564
- Single Agent Dose Level 3 (Experimental): Single Agent Dose Level 3
  Interventions: Drug: RNDO-564
- Single Agent Dose Level 4 (Experimental): Single Agent Dose Level 4
  Interventions: Drug: RNDO-564
- Single Agent Dose Level 5 (Experimental): Single Agent Dose Level 5
  Interventions: Drug: RNDO-564
- Single Agent Dose Level 6 (Experimental): Single Agent Dose Level 6
  Interventions: Drug: RNDO-564
- Single Agent Dose Level 7 (Experimental): Single Agent Dose Level 7
  Interventions: Drug: RNDO-564
- Single Agent Dose Level 8 (Experimental): Single Agent Dose Level 8
  Interventions: Drug: RNDO-564
- Single Agent Dose Level 9 (Experimental): Single Agent Dose Level 9
  Interventions: Drug: RNDO-564
- Combination Dose Escalation- Dose Level 1 (Experimental): Combination Dose Escalation- Dose Level 1
  Interventions: Drug: RNDO-564; Drug: Pembrolizumab
- Combination Dose Escalation - Dose Level 2 (Experimental): Combination Dose Escalation - Dose Level 2
  Interventions: Drug: RNDO-564; Drug: Pembrolizumab
- Single Agent Dose Optimization - Dose Level 1 (Experimental): Single Agent Dose Optimization - Dose Level 1
  Interventions: Drug: RNDO-564
- Single Agent Dose Optimization - Dose Level 2 (Experimental): Single Agent Dose Optimization - Dose Level 2
  Interventions: Drug: RNDO-564
- Combination Dose Optimization - Dose Level 1 (Experimental): Combination Dose Optimization - Dose Level 1
  Interventions: Drug: RNDO-564; Drug: Pembrolizumab
- Combination Dose Optimization- Dose Level 2 (Experimental): Combination Dose Optimization - Dose Level 2
  Interventions: Drug: RNDO-564; Drug: Pembrolizumab

INTERVENTIONS:
Drug: RNDO-564 — CD28 x Nectin-4 bispecific
Drug: Pembrolizumab — Anti-PD-1 therapy
  Arms: Combination Dose Escalation - Dose Level 2; Combination Dose Escalation- Dose Level 1; Combination Dose Optimization - Dose Level 1; Combination Dose Optimization- Dose Level 2

SUMMARY:
The main goal of this study is to evaluate how safe and tolerable RNDO-564 is and to identify the best dose of RNDO-564 as a single agent and in combination with pembrolizumab. The study is focused on participants with certain solid tumors that are in an advanced stage and have certain tumor makers. This will be done by measuring the side effects that participants experience and how severe they are. Additionally, the study will evaluate how RNDO-564 moves into, through, and out of the body and how the treatment affects the body.

The second goal of this study is to evaluate how well RNDO-564 works by itself or in combination with pembrolizumab at treating participants' cancer. This will be done by measuring the number of participants who respond to the treatment. The length of time where the tumor does not grow or spread will also be measured.

Participants will take RNDO-564 weekly on Days 1, 8 and 15 of a 21 day cycle. Participants in the combination arms will take RNDO-564 as described with pembrolizumab every 3 weeks.

DETAILED DESCRIPTION:
The study will consist of four stages: 1) single agent dose escalation, 2) single agent dose optimization, 3) combination dose escalation and 4) combination dose optimization.

Stages 1 and 3 are dose escalation to investigate the safety and tolerability of increasing doses of RNDO-564 as a single agent and in combination with standard pembrolizumab treatment. Participants will be enrolled who have one of the following advanced solid tumors associated with Nectin-4: locally advanced/metastatic urothelial cancer (la/m UC), cervical cancer (CC), head and neck cancer (HNSCC), esophageal cancer (EC), gastric (GC) and gastroesophageal junction cancer (GEJ), triple negative breast cancer (TNBC), and non-small cell lung cancer (NSCLC). The cancer must not have responded well to previous cancer treatments. Stages 1, and 3 will be non-randomized.

Stages 2 (i.e., RNDO-564 single agent) and 4 (i.e., RNDO-564 in combination with pembrolizumab) are dose optimization and proof-of-concept stages to further investigate the safety and tolerability of at least 2 doses of RNDO-564 as a single agent and in combination with standard pembrolizumab treatment, and to investigate preliminary anti-tumor activity. Stages 2 and 4 will enroll participants with advanced urothelial cancer only. The cancer must not have responded well to previous cancer treatments. Participants will be randomized (1:1) into one of two arms which will evaluate two dose levels (as selected from Stages 1 and 3).

The study consists of a screening period, a treatment period, an end of treatment visit, a safety follow-up visit, and 60 and 90 days telephone follow-up after ending treatment. The treatment period will last for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1) Eligible tumor types: Histologic documentation of incurable, locally advanced or metastatic solid tumors for which established standard systemic therapies are no longer effective (participant must have experienced progressive disease), are not tolerated, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds or have been declined by the participant, with these tumor subtypes:

A. Monotherapy and Combination Dose Escalation Arms:

* RR la/mUC: Participants with urothelial cancer (transitional cell) with squamous differentiation or mixed cell types are eligible. Participants with upper tract disease, e.g., involving ureters, or renal pelvis, are eligible. Participants may have had up to 2 prior monomethyl auristatin E (MMAE)-containing therapies, assuming any existing peripheral neuropathy is Grade 2 or less.
* NSCLC
* HNSCC
* CC
* GC and GEJ
* EC
* TNBC

B. Dose Optimization (Monotherapy and Combination Arms):

* Limited to participants who have RR la/mUC,
* Participants may have had up to 2 prior MMAE-containing therapies, assuming any existing peripheral neuropathy is Grade 2 or less 2. Participants must have measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1.

  3. Adequate organ function

Exclusion Criteria:

1. For Nectin-4 targeted agents (approved or investigational)

   * > one prior Nectin-4 targeted agents
2. Peripheral neuropathy > Grade 2
3. Participants with a history of, or with active, inflammatory skin disease, such as eczema, psoriasis that required or currently require biologics or oral steroids to control disease are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
All Arms: - Proportion of participants with adverse events (including dose limiting toxicities) as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 | From Day 1 to 90-days post last dose
  • Type, frequency, and severity of adverse events (AEs)
Dose Optimization Arms: • Identify one or more recommended Phase 2 doses (RP2D) | From Day 1 up to 24 months
  To evaluate the totality of data

SECONDARY OUTCOMES:
All Arms: To evaluate serum concentrations at specified timepoints of RNDO-564 as a single agent or in combination with pembrolizumab | From Day 1 up to 25 months (inclusive of 30 day safety follow-up)
All Arms: Proportion of participants that develop anti-drug antibodies to RNDO-564 | Baseline (predose) up to 25 months (inclusive of 30 day safety follow-up)
All Arms: Evaluate the prevalence, incidence and impact of anti-drug antibodies to RNDO-564 | From Baseline (predose) up to 25 months (inclusive of the 30 day safety follow-up).
All Arms: Objective Response Rate Among Participants | percentage of participants from Day 1 until the date of the first documented partial response or complete response assessed up to 24 months
All Arms: Duration of Response | Time between the first partial response or complete response and the date of first documented progression or date of death, whichever came first, assessed up to 24 months
All Arms: Median Progression Free Survival Time Among Participants | The number of months from Day 1 until the date of first documented progression or date of death, whichever came first, assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Manley, MD, Study Director — Rondo Therapeutics
Locations (2):
- United States (2):
  - Carolina Biooncology, Huntersville, North Carolina
  - Sarah Cannon Research Institute, LLD, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No